CLINICAL TRIAL: NCT04865380
Title: Does Tranexamic Acid Improve Visualization During Arthroscopic Rotator Cuff Repair: A Double Blinded, Randomized Control Trial
Brief Title: Does Tranexamic Acid Improve Visualization During Arthroscopic Rotator Cuff Repair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jeremy Reed, Principle Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-1983
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Subacromial Impingement; Subacromial Impingement Syndrome
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeons are blinded to group allocation and all treatment is administered by the anesthesia care provider. Patients will not be informed of their allocation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Tranexamic Acid (No Intervention): The anesthesiologist will not administer Tranexamic Acid at any point.
- Intravenous Tranexamic Acid (Experimental): 1g of Tranexamic Acid will be administered intravenously prior to the start of the operation.
  Interventions: Drug: Tranexamic Acid 100 MG/ML

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — 1g IV x 1 dose of Tranexamic Acid administered preoperatively.
  Other Names: Sandoz Tranexamic Acid Injection BP 100mg/mL, DIN 02246365
  Arms: Intravenous Tranexamic Acid

SUMMARY:
This clinical trial examines whether intravenous preoperative administration of tranexamic acid (TXA) before arthroscopic rotator cuff repair (ARCR) can improve arthroscopic visualization during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100
* Male and Female
* Patient able to read and understand consent form
* Non-traumatic, simple small or medium sized rotator cuff tear as defined by pre-operative MRI
* Booked to operating room for elective rotator cuff repair
* Beach chair positioning

Exclusion Criteria:

* Patient refusal to participate
* Massive rotator cuff tear
* Acute traumatic rotator cuff tear
* Known coagulopathy
* Patients with a history or risk of thromboembolism
* Known hypersensitivity to tranexamic acid
* Patient unable to be off anti-coagulant medication for long enough to counter effects
* Patient has a clinic systolic blood pressure > 150mmHg
* Lateral positioning
* Requirement or insistence by patient or anesthesiologist on regional block
* Patients who have smoked nicotine products within the last year
* The presence of other inflammatory conditions (calcific tendonitis, rheumatoid arthritis, etc.)
* The presence of active thromboembolic disease, such as deep vein thrombosis, pulmonary embolism, and cerebral thrombosis
* Patient has a seizure disorder
* Patients on medications identified as having drug-drug interactions (hormonal contraceptive, hydrochlorothiazide, desmopressin, sulbactam-ampicilllin, carbazochrome, ranitidine, or nitroglycerine
* Patient is pregnant
* Patients with history of subarachnoid hemorrhage
* Patients with renal insufficiency
* Patients with acquired disturbances of color vision

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Arthroscopic Visualization Score | Surgeon will complete the visualization score immediately after the surgery is completed.
  A visualization score from 1 to 6 assessed by the surgeon.
  1. - Perfect visualization
  2. - Mild difficulty that could easily be worked around
  3. - Moderate difficulty that required modifications to the surgical plan
  4. - Significant difficulty that added more than 10 minutes to the case
  5. - Major difficulty that added more than 20 minutes to the case
  6. - Difficulty that forced the stoppage of the case

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Reed, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Dash & Reed Sports Medicine, White City, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No